CLINICAL TRIAL: NCT00035022
Title: Phase I-II Study of Intravenous BCX-1777 in Relapsed or Refractory Aggressive (High Grade) T-Cell Malignancies
Brief Title: Study of Intravenous BCX-1777 in Relapsed or Refractory Aggressive T-Cell Leukemias or Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-01-02; NCT00066235 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-01-13 (Estimated); Status verified 2005-02

CONDITIONS: Leukemia, Lymphocytic; Lymphoma
Keywords: Leukemia, Lymphoma, T-Cell
MeSH Terms: conditions — Leukemia, Lymphoid; Lymphoma; Leukemia | interventions — forodesine

INTERVENTIONS:
Drug: BCX-1777

SUMMARY:
The purpose of this study is to determine if intravenous BCX-1777 can be given safely to improve relapsed or refractory aggressive T-cell leukemias and lymphomas.

DETAILED DESCRIPTION:
Despite the great strides that have been made in improving the outcome with frontline programs of intensive chemotherapy in patients with aggressive T-cell malignancies, the prognosis with relapsed or refractory T-cell leukemias or lymphomas is poor. BCX-1777 is a purine nucleoside phosphorylase (PNP) inhibitor and a potential T-cell target therapy.

The purpose of the phase I portion of the study is to determine the maximum tolerated dose (MTD) of BCX-1777 and the dose to be studied in the phase II portion of the study.

The purpose of the phase II portion of the study is to determine the safety and efficacy of BCX-1777 in patients with relapsed or refractory aggressive T-cell malignancies.

Patients who respond to BCX-1777 or have stable disease may be eligible to receive an additional course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated, relapsed or refractory aggressive T-cell malignancies (leukemias and lymphomas) histologically proven with measurable disease.
* Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
* All ages are eligible. Pediatric patients (<15 years of age) are eligible to be treated at a dose level previously tested in adults.
* Adequate liver and renal function.
* Patients with prior history of stem cell transplant if they meet all other eligibility requirements.
* Negative pregnancy test within 72 hours of study treatment in females of childbearing potential.
* Life expectancy of at least 2 months.

Exclusion:

* Active serious infection not controlled by oral or intravenous antibiotics.
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side-effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator.
* Concurrent treatment with other anti-cancer agents.
* Known CNS leukemia or lymphoma requiring intrathecal or craniospinal radiation therapy. Lumbar puncture not required in asymptomatic patients.
* Pregnant and/or lactating women; or fertile men or women not willing to use contraception.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71
Dates: Start 2001-08; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Thomas, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States